CLINICAL TRIAL: NCT05197205
Title: Nasopharyngeal Bacterial Carriage and Antibiotic Resistance in Children With Sickle Cell Disease in Ile-De-France
Acronym: DREPANO-BACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: APHP211360
Record Dates: First submitted 2021-12-09; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-10

CONDITIONS: Sickle Cell Disease
Keywords: Sickle celle disease, Nasopharyngeal bacterial carriage
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sickle cell children group (Experimental): A nasopharyngeal swab is taken during the consultation, with bacteriological analysis.
  Interventions: Procedure: nasopharyngeal swabbing
- control children group (No Intervention): healthy children control group (ACTIV network)

INTERVENTIONS:
Procedure: nasopharyngeal swabbing — A nasopharyngeal swab is collected during the consultation, with bacteriological analysis. No follow-up visit is required for this study
  Arms: sickle cell children group

SUMMARY:
The objective of this study is to to determine the rate of nasopharyngeal carriage of Streptococcus pneumoniae (Sp) in children with sickle cell disease over 6 months and under 15 years of age over a 9-month period in Ile-De-France.

DETAILED DESCRIPTION:
Sickle cell disease is the most common genetic disease in France, with one affected child for every 1,736 births. Ile-de-France is the region in Europe with the highest prevalence of sickle cell disease.

Children with sickle cell disease have an increased susceptibility to infections related to encapsulated bacteria and are at high risk of invasive infections (particularly Streptococcus pneumoniae), which is the leading cause of mortality in children with sickle cell disease under 5 years of age worldwide.

the patients are subject to intense selection pressure (long-term antibiotic prophylaxis and systematic probabilistic curative antibiotic therapy) and are at high risk of carrying nosocomial bacteria (repeated hospitalizations). Moreover, children with sickle cell disease have reinforced immunization schedules, especially against pneumococcal disease.

However, data concerning the carriage of resistant bacteria (prevalence, risk factors) in children with sickle cell disease in France are scarce.

This study aims to determine the nasopharyngeal bacterial carriage and antibiotic resistance in children with sickle cell disease in Ile-De-France

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to 15 years, regardless of immunization status.
* Child with a major sickle cell syndrome (SS, SC, S+, S°, SE) followed in one of the centers of competence or reference for rare diseases (CRMR) " Major sickle cell syndromes, Thalassemias and other rare pathologies of the Red Blood Cell and Erythropoiesis " in Ile de France.
* Children who are not subject to legal protection measures.
* Child affiliated to a social security system.
* Signed informed consent

Exclusion Criteria:

* Sickle cell child with a febrile syndrome at the time of sampling or hospitalized for any reason.
* Child having received antibiotic therapy other than oracillin in the 7 days preceding the nasopharyngeal swab.
* Child already included in the observation period (only 1 nasopharyngeal swab per patient).
* Other hemoglobinopathies and heterozygous AS or AC patients.
* Patients already involved in a therapeutic protocol or in the exclusion period following a previous research.
* Patients under AME or without social security coverage.

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
determine the proportion of sickle cell children with nasopharyngeal carriage of Streptococcus pneumoniae (Sp) among the total number of sickle cell children screened by nasopharyngeal swab. | 12 months
  the rate of nasopharyngeal carriage of Streptococcus pneumoniae (Sp) in children with sickle cell disease aged over 6 months and under 15 years over a 12-month period in Ile-De-France.

SECONDARY OUTCOMES:
determine the rate of nasopharyngeal carriage of penicillin-deficient pneumococcus (PDSP) in sickle cell children over 6 months and under 15 years of age over a 9-month period in Ile-De-France. | 12 months
  Proportion of sickle cell children with nasopharyngeal carriage of penicillin-deficient pneumococcus (PDSP) among the total number of sickle cell children screened by nasopharyngeal swab.
determine the proportion of vaccine serotypes among pneumococcal strains in children with sickle cell disease aged over 6 months and under 15 | 12 months
  Proportion of children with vaccine serotypes among the pneumococcal strains
Determine the proportion of non-vaccine serotypes among all pneumococcal strains in children with sickle cell disease over 6 months and under 15 years of age. | 12 months
  Proportion of non-vaccine serotypes among all pneumococcal strains.
Determine the nasopharyngeal carriage rate of methicillin-resistant Staphylococcus aureus (MRSA), Haemophilus influenzae, Moraxella catarrhalis in children with sickle cell disease over 6 months and under 15 years of age. | 12 months
  Proportion of children with MRSA, Haemophilus influenzae, Moraxella Catarrhalis (isolated from a nasopharyngeal swab).
compare the rate of nasopharyngeal carriage of Streptococcus pneumoniae and PSDP between the sickle cell group and the healthy group of children according to age groups. | 12 months
  Proportion of children with Streptococcus pneumoniae and PSDP (isolated on nasopharyngeal swab) by age group.
Compare the proportion of non-vaccine serotypes among the Streptococcus pneumoniae strains between the sickle cell group and the healthy group of children. | 12 months
  Proportion of non-vaccine serotypes among nasopharyngeal strains of Streptococcus pneumoniae.
compare the nasopharyngeal carriage rate of MRSA, Haemophilus influenzae, Moraxella catarrhalis between the sickle cell group and the healthy children group. | 12 months
  Proportion of children with MRSA, Haemophilus influenzae, Moraxella Catarrhalis (isolated on nasopharyngeal swab).

REFERENCES:
- [Background] Schaumburg F, Biallas B, Ngoune Feugap E, Alabi AS, Mordmuller B, Kremsner PG, Grobusch MP, Lell B, van der Linden M, Peters G, Adegnika AA. Carriage of encapsulated bacteria in Gabonese children with sickle cell anaemia. Clin Microbiol Infect. 2013 Mar;19(3):235-41. doi: 10.1111/j.1469-0691.2012.03771.x. Epub 2012 Feb 13. PMID 22329610
- [Background] Dayie NTKD, Tetteh-Ocloo G, Labi AK, Olayemi E, Slotved HC, Lartey M, Donkor ES. Pneumococcal carriage among sickle cell disease patients in Accra, Ghana: Risk factors, serotypes and antibiotic resistance. PLoS One. 2018 Nov 8;13(11):e0206728. doi: 10.1371/journal.pone.0206728. eCollection 2018. PMID 30408061
- [Background] Schaumburg F, Biallas B, Alabi AS, Grobusch MP, Feugap EN, Lell B, Mellmann A, Peters G, Kremsner PG, Becker K, Adegnika AA. Clonal structure of Staphylococcus aureus colonizing children with sickle cell anaemia and healthy controls. Epidemiol Infect. 2013 Aug;141(8):1717-20. doi: 10.1017/S0950268812002270. Epub 2012 Oct 10. PMID 23050673
- [Derived] Pham LL, Varon E, Bonacorsi S, Boubaya M, Benhaim P, Amor-Chelihi L, Houlier M, Koehl B, Missud F, Brousse V, Gajdos V, Bizot E, Briand C, Malka A, Odievre MH, Romain AS, Hau I, Pondarre C, See H, Guitton C, Zenkhri F, Holvoet L, Benkerrou M, Da Silveira C, Belaid N, Laurent O, Vassal M, Basmaci R, Aupiais C, Bloch-Queyrat C, Levy C, Cohen R, Ouldali N, De Pontual L, Carbonnelle E, Gaschignard J. Nasopharyngeal Carriage and Antibiotic Resistance in Children With Sickle Cell Disease: The DREPANOBACT French Multicenter Prospective Study. Pediatr Infect Dis J. 2025 May 1;44(5):387-393. doi: 10.1097/INF.0000000000004744. Epub 2025 Feb 3. PMID 40232881